CLINICAL TRIAL: NCT04357028
Title: Effectiveness of Measles Vaccine in Health Care Professionals During COVID-19 Outbreak (Randomized Controlled Trial)
Brief Title: Measles Vaccine in HCW
Acronym: MV-COVID19
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Failure of subject recruitment
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mukhtar, professor of anesthesia and intensive care, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N-30-2020
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: MMR vaccine, Respiratory failure,
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMR vaccine (Experimental): 0.5 ml subcutaneous of MMR vaccine will be injected in posterior triceps aspect of upper arm
  Interventions: Drug: Measles-Mumps-Rubella Vaccine
- Control (Placebo Comparator): 0.5 ml subcutaneous of saline will be injected in posterior triceps aspect of upper arm
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Measles-Mumps-Rubella Vaccine — Measles mumps Rubella vaccine is a weak attenuated life vaccine
  Arms: MMR vaccine
Drug: Placebos — 0.5 ml subcutaneous of saline will be injected in posterior triceps aspect of upper arm
  Arms: Control

SUMMARY:
Till now, mortality reports among children below 9 years remains extremely low despite that the incidence of death toll is high and exceeding 50,000 patients among older population, One speculation for lower SARS infectivity is that cross-protective antibodies against measles vaccine ( MV). In mice susceptible to measles virus, recombinant MV induced the highest titers of neutralizing antibodies and fully protected immunized animals from intranasal infectious challenge with SARS-CoV,

The primary objective of the present study is to determine the benefit of measles vaccine in health care professional to decrease the incidence of COVID-19.

We Hypothesized that, measles vaccine may lower the incidence of serologically proven SARS-CoV-2 infection and reported respiratory illness

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years old
* Subjects who are willing to comply with the requirements of the study protocol and scheduled visits (for example, completion of the subject diary, return for follow-up visits) and who are willing to make themselves available for the duration of the study with access to a consistent means of telephone contact

Exclusion Criteria:

* acute severe illness
* recent receipt of a blood product
* history of thrombocytopenia
* Pregnant females
* any chronic medical condition
* Any participant receiving any immune suppressive medication
* Immunocompromised staff
* Participants who have egg allergy
* Participants who care for immune compromised hosts
* Participants who test positive for COVID-19 serology prior to randomization

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
COVID-19 disease incidence | Time Frame: Measured over the 6 months following randomization
  Number of participants with asymptomatic or mild COVID-19 disease defined as fever (using self-reported questionnaire), plus at least one sign or symptom of respiratory disease including cough, runny/blocked nose (using self-reported questionnaire), plus positive SARS-Cov-2 test (PCR or serology)

SECONDARY OUTCOMES:
SARS-CoV-2 pneumonia | Time Frame: Measured over the 6 months following randomization
  Number of pneumonia cases (abnormal chest X-ray) (using self-reported questionnaire and/or medical/hospital records) associated with a positive SARS-CoV-2 test
Critical care admission duration with SARS-CoV-2 | Time Frame: Measured over the 6 months following randomization
  Number of days admitted to critical care (using self-reported questionnaire and/or medical/hospital records) associated with a positive SARS-CoV-2 test
Oxygen therapy with SARS-CoV-2 | Time Frame: Measured over the 6 months following randomization
  Need for oxygen therapy (using self-reported questionnaire and/or medical/hospital records) associated with a positive SARS-CoV-2 test

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No